CLINICAL TRIAL: NCT04914455
Title: Performance of Static and Dynamic Accessment of Inferior Vena Cava Diameter for the Diagnosis of Fluid Responsiveness
Brief Title: Transhepatic Echography for Fluid Responsiveness After Cardiovascular Surgery
Acronym: THEFRACS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_17; 2019_17 2019-A02724-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Inferior Vena Cava Abnormality; Fluid Responsiveness; Fluid Overload; Venous Congestion; Cardiovascular Surgery
Keywords: Inferior vena cava distensibility; Transhepatic inferior vena cava distensibility; Ultrasound diagnoses
MeSH Terms: conditions — Edema; Hyperemia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fluid responsiveness groups (responders and non-responders): Fluid responsiveness is defined as an increase in stroke volume of 10% and more form baseline.
  Interventions: Diagnostic Test: Echocardiography and transhepatic inferior vena cava assessment using ultrasound.

INTERVENTIONS:
Diagnostic Test: Echocardiography and transhepatic inferior vena cava assessment using ultrasound. — For all participant :
  * Inferior vena cava diameter will be measure before and after fluid expansion 'which administration will be decided by a physician other that the investigator).
  * Stroke volume using primarily VTI in TTE or a cardiac output monitoring device (Swan ganz catheter (Edwards life science), EV 1000 (edwards life science), PiCCO(Getinge))
  * Absence of significant pericardial effusion of hematoma
  Whenever possible:
  Subcostal measurement of IVC, ejection fraction, cardiac outcput, mitral E, A and E' waves, TAPSE, tricupid S' wave, Right ventricle fractional area change.
  venous congestion assesment : hepatic vein, portal vein and renal vein Doppler to define the VEXUS Score;
  Other Names: Venous congestion using ultrasound

SUMMARY:
Fluid expansion in critically ill patients following high risk surgery may induce fluid overload and worse outcome. Several tools have been developped to predict fluid responsiveness in such situation in order to avoid inappropriate fluid administration but with several limitations. Inferior vena cava (IVC) distensibility is one of those tools which has the advantage to be non-invasive, dynamic and safe, is usually measured by subcostal (SC)approach. In post surgical setting this acess is limited du to practical reasons (scar, dressing...), therefore a transhepatic (TH) approach is used but has not been validated as a fluid responsiveness prediction tool. The correlation between SC approach with the TH approach vary according to studies. Therefore the performances, the threshold identified for SC approach can not be translated to the TH approach. Further, fluid congestion status measured before IVC analyses, may be a useful confounder and safety endpoint for fluid responsiveness interpretation.

The primary objective of this study is therefore to study the performance of the IVC measured using TH approach (IVCth) in predicting of fluid responsiveness defined as an increased of 10% and over of stroke volume.

Secondary objectives intend to analyse the correlation between TH and SC approaches, to compared their performances for fluid responsiveness prediction, and to analyse the weight of venous congestion on fluid responsiveness prediction.

DETAILED DESCRIPTION:
Inappropriate volume expansion in the critically ill patient may leads to an increase in fluid balance, fluid overload and worse outcome. This increase in fluid balance is associated with a poor prognosis in the ICU patients, especially after cardiac surgery and high risk surgery .

Generally, the primary objective of an adequate volume expansion is a significant increase in stroke volume called fluid responsiveness (> 10% of increase). This increase in cardiac output promotes tissue perfusion, thus avoiding the occurrence of organ dysfunction.

The identification of fluid responsiveness in these patients is thus a cardinal element of haemodynamic management in intensive care. Among the non-invasive tools to assess this fluid responsiveness, the assessment of the ventilatory or forced inspiration distensibility of the inferior vena cava (IVC) has been proposed with convincing results in several clinical studies. However with various diagnostic performances and threshold.

The measurement of the diameter of the IVC is classically performed via the subcostal (SC) or subxiphoid approach. However, this approach is not always easily accessible in intensive care patients, particularly after cardiovascular surgery or laparotomy, due to practical constraints (algic scars, dressings, prone position). The transhepatic approach (TH) is a technically feasible approach in such cases. However, it has little validation in the literature, particularly in its ability to predict response to volume expansion. knowing that the correlation between the SC approach with the TH approach varies according to studies, the performance and the threshold identified for SC approach can not be translated into that of the TH approach. Further, fluid congestion status measured before IVC analyses, may be a useful confounder and safety endpoint for fluid responsiveness interpretation.

ELIGIBILITY:
Inclusion Criteria:

* High risk cardiovascular surgery patients admitted in ICU
* With transhepatic IVC and stroke volume measurement feasible.
* Informed consent

Exclusion Criteria:

* Righ ventricle failure
* Significant tricuspid regurgitation
* Tamponade
* Severe hypoxemia
* Age <18 ans
* No health care coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our intensive care unit following cardiac surgery or aortic surgery, under mechanical ventilation or not.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | Measurement performs before and after fluid bolus (during the 10 min following the end of fluid bolus).
  An increase in stroke volume of 10% and more, following fluid bolus of 250 to 500 ml of cristalloid or colloid.

SECONDARY OUTCOMES:
Venous congestion | during the 15 minutes following the end of the fluid bolus
  Venous congestion is defined using the VEXUS Score after sub hepatic, portal and renal veins Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Mouhamed MOUSSA, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service d'Anesthésie-Réanimation CCV Hôpital Cardiologique Centre Hospitalier et Universitaire de Lille, Lille, NORD, France